CLINICAL TRIAL: NCT05382624
Title: The Relationship Between Abdominal Circumference: Hip Ratio and Ephedrine Requirement in Spinal Anesthesia for Elective Cesarean: A Prospective Observational Study
Brief Title: The Relationship Between Abdominal Circumference: Hip Ratio and Ephedrine Requirement
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet AKSOY, Assoc. Prof. Dr., Ataturk University
Other Study IDs: BEAH KAEK 2021/05-100
Record Dates: First submitted 2022-05-07; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hypotension; Anesthesia, Local; Cesarean Section Complications
Keywords: hypotension; spinal anesthesia; cesarean section; ephedrine requirement; abdominal circumference; hip circumference,
MeSH Terms: conditions — Hypotension | interventions — Anesthesia, Spinal; Postoperative Period

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing cesarean with spinal anesthesia: The AC-to-hip ratio was calculated by dividing the values of the abdominal (cm) and hip circumference (cm). Spinal anesthesia in the sitting position was performed in all patients using 2.4 ml 0.5% hyperbaric bupivacaine (12 mg). Intravenous ephedrine (5 mg) was given in case of persistent hypotension. The number of patients requiring ephedrine and the total amount of ephedrine used during surgery were recorded.
  Interventions: Procedure: Abdominal circumference was measured at the umbilical level in the standing position at the end of a normal expiration.

INTERVENTIONS:
Procedure: Abdominal circumference was measured at the umbilical level in the standing position at the end of a normal expiration. — The operation time (the time from the beginning of the surgical incision until the end of surgery), anesthetic complications, such as nausea or vomiting, the number of patients requiring ephedrine and atropine, the total amount of intravenous fluid used, and the total amount of ephedrine used during surgery were recorded.
  Other Names: Hip circumference was measured at the widest circumference over the buttocks.; Three consecutive measurements were obtained; results were averaged and the AC-to-hip ratio was calculated by dividing the values of the abdominal (cm) and hip circumference (cm).; Spinal anesthesia in the sitting position was performed on all patients.; After surgery, patients were transferred to the recovery room.

SUMMARY:
This prospective observational study aimed to investigate whether there is a relationship between weight, height, BMI, abdominal circumference (AC), hip circumference (HC), and AC-to-hip ratio with the incidence of hypotension in patients undergoing cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
This prospective observational study was conducted over eight months from March 2021 to October 2021 at the Anesthesiology and Reanimation Department of Erzurum Regional Training and Research Hospital, Erzurum, Turkey, a tertiary care hospital. Before commencing the study, the Institute ethics committee approval was taken from the Ethical Committee of Health Sciences University, Erzurum Regional Training and Research Hospital, Erzurum, Turkey. This study was carried out in accordance with the Declaration of Helsinki and written informed consent was obtained from all participants.

The study population comprised 60 women who agreed to participate with uncomplicated term pregnancies, BMI < 30 kg/m2, aged between 18-45 years, ASA I and II undergoing elective cesarean section under spinal anesthesia. Participants with a complicated pregnancy, such as diabetes, hypertension, fetal anomaly, a history of allergy to study drugs, psychiatric diseases, coagulation abnormalities, and mul¬tiple pregnancies were excluded from the study. Also, patients who required conversion to general anesthesia were excluded.

A day before surgery, patients were informed about the study, and written informed consent was obtained from participants. On the day of the operation, all participants were preloaded with 500 milliliters of Ringer's lactate through a 16-18 gauge intravenous cannula. In the operating room, standard monitorization including non-invasive blood pressure, electrocardiography, and pulse oximetry was provided. Before the spinal anesthesia, patients' age, weight, height, abdominal and hip circumferences, ASA physical status, baseline values of noninvasive blood pressure, and heart rate (HR) were recorded.

Abdominal circumference was measured at the umbilical level in the standing position at the end of a normal expiration. Hip circumference was measured at the widest circumference over the buttocks. All the measurements were carried out by the trained anesthesia technician using standard non-stretch tape with the parturients wearing light clothes. To minimize errors, three consecutive measurements were obtained; results were averaged and the AC-to-hip ratio was calculated by dividing the values of the abdominal (cm) and hip circumference (cm).

Spinal anesthesia in the sitting position was performed on all patients. Following skin sterilization, a 27-gauge Quincke-tip spinal needle was advanced through the midline L3-4 intervertebral space. After free cerebrospinal fluid flow was observed, 2.4 ml 0.5% hyperbaric bupivacaine (12 mg) was injected over 30 seconds. Then, the spinal needle was removed and patients were placed in the supine position for the operation, and the operating table was tilted 20° to the left. A pinprick test was used to evaluate the sensory block level and surgery was initiated when the sensory block reached the T6 dermatome. Spinal anesthesia was considered to have failed when the sensory block was not consistent within the first 20 minutes following the spinal injection. In this instance, general anesthesia was performed and these patients were excluded from the study. A Modified Bromage scale was used to evaluate the motor block level. After delivery of the baby, 20 IU oxytocin in 1000 ml Ringer's lactate solution was given intravenously over 5 hours. Hypotension (a 20% decrease in systolic blood pressure compared to preoperative values), was treated by uterine displacement and rapid infusion of fluid. Intravenous ephedrine (5 mg) was given in case of persistent hypotension. Intravenous atropine (1 mg) was injected to treat bradycardia (the HR < 45 beats/minute). In our clinic, ephedrine is routinely used as the first choice in the treatment of hypotension. Intravenous ondansetron (4 mg) was used to treat persistent nausea and vomiting. Following spinal injection, systolic, diastolic, and mean arterial pressure and HR values were recorded every 2 minutes for 20 minutes and then every 5 minutes until the end of the operation. The operation time (the time from the beginning of the surgical incision until the end of surgery), anesthetic complications, such as nausea or vomiting, the number of patients requiring ephedrine and atropine, the total amount of intravenous fluid used, and the total amount of ephedrine used during surgery were recorded. Neonatal Apgar scores at 1 and 5 minutes after delivery and the weight and height of the neonates were recorded. After surgery, patients were transferred to the recovery room. Pain severity was assessed via the Visual analog scale (VAS, 0 cm=no pain, 10 cm=worst pain). In the case of VAS > 3, 1 gr paracetamol was given to patients intravenously. Anesthesia-related side effects (e.g., nausea, vomiting, and headache), sensory block time (from the spinal injection to the recovery of T10 dermatome), and the time requiring supplemental analgesics was recorded by an independent observer blinded to the group assignment at 30 min and 1st and 2nd hours post-operatively. When the motor block had regressed to the T10 level, patients were sent to the clinics.

Statistical Analysis The sample size calculation was performed based on the data gained from the study's preliminary results using Russ Lenth's power and sample size calculation application (13). Fifty-eight patients were needed to detect an anticipated effect size of 0.37 with a power of 85% and an alpha of 5%.

The statistical analysis of all data was performed with SPSS 20 software (SPSS Inc., Chicago, IL, USA), and P<0.05 was considered statistically significant. Data were expressed as mean values ± standard deviation (SD), median (min-max), or number and percentage values. Kolmogorov-Smirnov test was used to detect the distribution of data.

Pearson correlation analysis was performed to assess the association between anthropometric measures (i.e., BMI, AC-to-hip ratio) with the incidence of hypotension and the total amount of ephedrine used. Correlation analysis was performed to find the correlations between the total amount of ephedrine used and the AC, HC, and AC-to-hip ratio. The correlation between the total amount of ephedrine used and the weight of the fetus was also investigated. The regression equations were obtained by using the linear regression method and the coefficients (r2) were compared.

ELIGIBILITY:
Inclusion Criteria:

* women who agreed to participate
* with uncomplicated term pregnancies
* BMI < 30 kg/m2
* aged between 18-45 years
* ASA I and II
* undergoing elective cesarean section under spinal anesthesia

Exclusion Criteria:

* a complicated pregnancy, such as diabetes, hypertension, fetal anomaly
* a history of allergy to study drugs
* psychiatric diseases
* coagulation abnormalities
* multiple pregnancies
* patients who required conversion to general anesthesia

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — women with uncomplicated term pregnancy
Study Population: The study population comprised 60 women who agreed to participate with uncomplicated term pregnancies, BMI < 30 kg/m2, aged between 18-45 years, ASA I and II undergoing elective cesarean section under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Ephedrine requirement | Two hours.
  Ephedrine requirement (mg) from the beginning to the end of the surgery.

SECONDARY OUTCOMES:
atropine requirement | Two hours.
  Atropine requirement (mg) from the beginning to the end of the surgery.
Blood pressure values | Baseline, during surgery.
  The change in systolic and diastolic blood pressure values (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah CAN, MD, Principal Investigator — Erzurum Regional Training and Research Hospital; Ayse N DAS, MD, Principal Investigator — Erzurum Regional Training and Research Hospital
Locations (1):
- Mehmet Aksoy, Erzurum, string:Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No